CLINICAL TRIAL: NCT03907410
Title: The Tailored Adherence Incentives for Childhood Asthma Medications (TAICAM) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 18-015434; 1K23HL136842-01A1 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Medication Adherence; Asthma in Children
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Incentives, plus reminders & feedback (IRF) (Experimental): There will be a run-in period to determine eligibility for randomization and collect baseline adherence data (Month 0).
  During the "Experiment" period (Months 1-3), Arm 1 will receive the IRF intervention.
  During the "Observation" period (Months 4-6), all the arms will have continued daily ICS monitoring to assess enduring effects of each arm - no IRF.
  Interventions: Other: Nominal Financial Incentives; Other: Daily Adherence Reminders/Adherence Performance Feedback
- Arm 2: Reminders & feedback ONLY (Active Comparator): There will be a run-in period to determine eligibility for randomization and collect baseline adherence data (Month 0).
  During the "Experiment" period (Months 1-3), Arm 2 will receive ONLY reminders and feedback, without nominal financial incentives.
  During the "Observation" period (Months 4-6), all three arms will have continued daily ICS monitoring to assess enduring effects of each arm - no IRF.
  Interventions: Other: Daily Adherence Reminders/Adherence Performance Feedback
- Arm 3 (Control) (No Intervention): There will be a run-in period to determine eligibility for randomization and collect baseline adherence data (Month 0).
  During the "Experiment" period (Months 1-3), Arm 3 will not receive any component of the IRF intervention.
  During the "Observation" period (Months 4-6), all three arms will have continued daily ICS monitoring to assess enduring effects of each arm - no IRF.

INTERVENTIONS:
Other: Nominal Financial Incentives — The nominal financial incentives will consist of fixed-ratio incentives for each inhaled corticosteroids (ICS) actuation (25 cents for children on 4 daily ICS doses and 50 cents for children on 2 daily doses), with a maximum of $1 per day.
  Arms: Arm 1: Incentives, plus reminders & feedback (IRF)
Other: Daily Adherence Reminders/Adherence Performance Feedback — Study participants will receive automated daily text message or push notification reminders and automated weekly feedback summarizing their adherence performance through Way to Health, a mobile health, electronic monitoring platform.
  Arms: Arm 1: Incentives, plus reminders & feedback (IRF); Arm 2: Reminders & feedback ONLY

SUMMARY:
Improving adherence to inhaled corticosteroids (ICS) medication in urban minority pediatric populations is a clinical and population health priority. Financial incentives have been shown as a compelling method to engage a high-risk asthma population in regular ICS use, but whether and how adherence can be maintained and lead to sustained high adherence trajectories is unknown.

DETAILED DESCRIPTION:
Investigators propose to initially enroll 125 children into an initial 1-month run-in interval. Participants who successfully complete the run-in interval will be randomized into a six-month intervention with a six month follow-up period. Children will be ages 5-12, and must have two or more visits to any combination of the outpatient, Emergency Department (ED) or hospital setting in the past year for asthma exacerbations at Children's Hospital of Philadelphia (CHOP).

The study intervention will include daily automated medication reminders (either via text message or push reminder), an app to track daily medication use, and nominal incentives to promote daily controller use. Inhaled controller medication adherence and rescue medication use will be measured using electronic monitors affixed to the inhalers. Factors associated with differential adherence will be assessed using surveys administered during enrollment, the experiment interval (months 1 through 3), the observation interval (months 4 through 6), and study completion (months 12-13). Efficacy outcomes will include change in parent-reported asthma control and mean adherence to ICS between study arms during the experiment interval, as well as the observation interval.

Patients will be considered fully enrolled when they fulfill the requirements of the Run-in period (sensor data uploaded to research platform AND text message receipt confirmed by caregiver) and are subsequently randomized.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 5 to 12 years and their parent or legal guardian.
* Caregiver has an app enabled cellular phone (i.e., smart phone)
* Prescribed inhaled corticosteroid or corticosteroid/long acting beta agonist combination for daily use
* At least 2 asthma exacerbations in the preceding year (Any combination of hospitalizations, ED visits, or outpatient visits where oral steroid courses were administered for asthma)
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

* Subjects prescribed a controller medication to which the electronic device cannot affix
* Subjects in which the mobile app is not compatible with their smart phone model
* Subjects with major developmental delays or disabilities
* Subjects with comorbid chronic diagnoses that influence their asthma management such as cystic fibrosis, bronchopulmonary dysplasia, or cyanotic heart disease
* Families with active Department of Human Services (DHS) involvement
* Non-English speaking families
* Parents/guardians or subjects whose medical team recommends against approaching for enrollment in a research study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Kenyon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenyon CC, Quarshie WO, Xiao R, Yazdani M, Flaherty CM, Floyd GC, Miller VA, Bryant-Stephens TC, Zorc JJ, Feudtner C. Tailored Adherence Incentives for Childhood Asthma Medications: A Randomized Clinical Trial. JAMA Pediatr. 2025 May 1;179(5):500-507. doi: 10.1001/jamapediatrics.2025.0010. PMID 40094638
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614
- [Derived] Henderson BR, Flaherty CM, Floyd GC, You J, Xiao R, Bryant-Stephens TC, Miller VA, Feudtner C, Kenyon CC. Tailored Medication Adherence Incentives Using mHealth for Children With High-Risk Asthma (TAICAM): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Aug 17;9(8):e16711. doi: 10.2196/16711. PMID 32459653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 125 participants were initially enrolled into the 1 month study run-in period, in which they were needed to successfully (1) synchronize their electronic study sensor with the caregivers smartphone (via Bluetooth) and the Way to Health study platform (via wireless or cellular data) and (2) respond to an automated text message from the Way to Health study platform.
Pre-assignment Details: 19 participants did not successfully complete the run-in period and, thus, were not randomized. 106 study participants were randomized in a 2:1:2 schema. The caregiver-child dyad was one unit. If the caregiver withdrew from the study, the child also withdrew from the study. Medication adherence was only collected from the child, but caregivers were included in the dyad-language given that they were interacting with certain parts of the intervention employed.
Groups:
- Arm 1: Incentives, Plus Reminders & Feedback (IRF): There will be a run-in period to determine eligibility for randomization and collect baseline adherence data (Month 0).
  During the "Experiment" period (Months 1-3), Arm 1 will receive the IRF intervention.
  During the "Observation" period (Months 4-6), all the arms will have continued daily ICS monitoring to assess enduring effects of each arm - no IRF.
  Nominal Financial Incentives: The nominal financial incentives will consist of fixed-ratio incentives for each inhaled corticosteroids (ICS) actuation (25 cents for children on 4 daily ICS doses and 50 cents for children on 2 daily doses), with a maximum of $1 per day.
  Daily Adherence Reminders/Adherence Performance Feedback: Study participants will receive automated daily text message or push notification reminders and automated weekly feedback summarizing their adherence performance through Way to Health, a mobile health, electronic monitoring platform.
- Arm 2: Reminders & Feedback ONLY: There will be a run-in period to determine eligibility for randomization and collect baseline adherence data (Month 0).
  During the "Experiment" period (Months 1-3), Arm 2 will receive ONLY reminders and feedback, without nominal financial incentives.
  During the "Observation" period (Months 4-6), all three arms will have continued daily ICS monitoring to assess enduring effects of each arm - no IRF.
  Daily Adherence Reminders/Adherence Performance Feedback: Study participants will receive automated daily text message or push notification reminders and automated weekly feedback summarizing their adherence performance through Way to Health, a mobile health, electronic monitoring platform.
Period: Overall Study
Arm/Group | Arm 1: Incentives, Plus Reminders & Feedback (IRF) | Arm 2: Reminders & Feedback ONLY | Arm 3 (Control)
Started | 42 | 22 | 42
Completed | 38 | 21 | 40
Not Completed | 4 | 1 | 2
Not completed — Lost to Follow-up | 4 | 1 | 1
Not completed — Lost to follow-up and research burden | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The "Sex (Female, Male)" and "Race/Ethnicity, Customized" baseline characteristics for the child were collected from the parent/caregivers involved in the study. These variables were not collected for the parents/caregivers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Incentives, Plus Reminders & Feedback (IRF) | Arm 2: Reminders & Feedback ONLY | Arm 3 (Control) | Total
Number analyzed (Participants) | 38 | 21 | 40 | 99
Age, Customized [Count of Participants; unit: Participants]
  Child Age Group: 5-7 years | 12 | 10 | 18 | 40
  Child Age Group: 8-11 years | 26 | 11 | 22 | 59
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean Caregiver Age | 34.2 (5.9) | 34.1 (5.6) | 33.5 (6.7) | 33.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Child Sex: Female | 18 | 9 | 16 | 43
  Child Sex: Male | 20 | 12 | 24 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Child Race: Black | 31 | 17 | 33 | 81
  Child Race: Non-Black | 7 | 4 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 38 | 21 | 40 | 99
Run-in Period ICS Adherence [Mean (Standard Deviation); unit: % of doses taken] | 56 (26) | 50 (29) | 52 (30) | 53 (28)

OUTCOME MEASURES:

1. Primary Outcome: Mean Monthly Adherence to Inhaled Corticosteroid Regimen (Unadjusted)
Description: Calculated as the mean daily proportion of prescribed doses taken by study month by study arm. Days that reflect >1 were truncated to 1.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: proportion of prescribed doses taken
Groups:
- Arm 1: Full intervention group
- Arm 2: Hybrid intervention group
- Arm 3: Active control group
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 38 | 21 | 40
proportion of prescribed doses taken
  Month 0 | 0.56 [0.52 to 0.61] | 0.50 [0.44 to 0.57] | 0.52 [0.47 to 0.57]
  Month 1 | 0.61 [0.57 to 0.66] | 0.48 [0.41 to 0.54] | 0.47 [0.41 to 0.52]
  Month 2 | 0.56 [0.52 to 0.61] | 0.45 [0.38 to 0.51] | 0.38 [0.33 to 0.43]
  Month 3 | 0.55 [0.49 to 0.60] | 0.44 [0.37 to 0.51] | 0.39 [0.34 to 0.45]
  Month 4 | 0.44 [0.39 to 0.48] | 0.40 [0.32 to 0.47] | 0.45 [0.39 to 0.50]
  Month 5 | 0.35 [0.29 to 0.40] | 0.30 [0.23 to 0.37] | 0.41 [0.35 to 0.46]
  Month 6 | 0.38 [0.34 to 0.42] | 0.34 [0.28 to 0.40] | 0.48 [0.43 to 0.53]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Multivariate comparison of Experiment phase adherence (Months 1-3) comparing Arm 1 (Full Intervention arm) to Arm 3 (Active control). Arm 3 is used as the reference. This randomized controlled trial was powered for Arm 1 vs. Arm 3 comparisons, hence the Arm 1 vs. Arm 3 outcome data for adherence to the inhaled corticosteroid regime. The study did not have sufficient power for Arm 2 comparisons; Test type: Superiority; Mean Difference (Final Values) = 15, 95% CI 2-sided [2 to 28]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 3; Multivariate comparison of Observation phase adherence (Months 4-6) comparing Arm 1 (Full Intervention arm) to Arm 3 (Active control). Arm 3 is used as the reference. This randomized controlled trial was powered for Arm 1 vs. Arm 3 comparisons, hence the Arm 1 vs. Arm 3 outcome data for adherence to the inhaled corticosteroid regime. The study did not have sufficient power for Arm 2 comparisons; Test type: Superiority; Mean Difference (Final Values) = -6, 95% CI 2-sided [-20 to 7]

2. Secondary Outcome: Adherence Trajectory
Description: Group-based trajectory modeling derived of adherence patterns - not reported by study arm. This secondary outcome was included in the event that there was no difference in adherence between study arms to help identify participant characteristics that were associated with different adherence patterns. The unit of measure is the percentage of participants that fall into each adherence category (low, medium, and high adherence) over a 6-month time period.
Time Frame: 6 months
Population: The total cohort of 99 participants were analyzed to assign participants to one adherence group based on their adherence to the inhaled corticosteroid medication over the study interval. As pre-specified in the study protocol, this outcome measure represents group-based modeling of adherence patterns agnostic of study arm.
Measure: Number; unit: percentage of study participants
Groups:
- Low Adherence: Percentage of participants with low adherence to their inhaled corticosteroid medication regimen
- Medium Adherence: Percentage of participants with medium adherence to their inhaled corticosteroid medication regimen
- High Adherence: Percentage of participants with high adherence to their inhaled corticosteroid medication regimen
Arm/Group | Low Adherence | Medium Adherence | High Adherence
Number analyzed (Participants) | 99 | 99 | 99
percentage of study participants | 20.2 | 41.5 | 38.2

3. Secondary Outcome: Changes in Child Asthma Control Tool (cACT) Score
Description: Assess the change in total cACT score or parental portion of the cACT from baseline to the second, third, fourth, and fifth study visits. The Child Asthma Control Tool (cACT) score ranges from 0 (poor control) to 27 (complete control) and was assessed at study visits 1 and 3 only. The parental portion of the cACT ranges from 0-15 and was assessed at all study visits. The greater the value, the better the control. The larger the difference (larger magnitude) of the value in the differences between the scores, the greater the improvement in controlling the child's asthma diagnosis.
Time Frame: months 2, 4,7, 12
Population: The number analyzed in the study visits differ as some participants did not complete all study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 1: Full Intervention
- Arm 2: Hybrid Intervention
- Arm 3: Active Control
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 38 | 21 | 40
score on a scale
  Study Visit 2* (only parental portion of ACT collected: Range 0-15) - Month 2: number analyzed (Participants) | 36 | 15 | 34
  Study Visit 2* (only parental portion of ACT collected: Range 0-15) - Month 2 | 1.73 (0.64) | 2.86 (0.73) | 2.16 (0.71)
  Study Visit 3 - Month 4: number analyzed (Participants) | 32 | 15 | 31
  Study Visit 3 - Month 4 | 2.19 (0.96) | 3.63 (1.15) | 1.85 (1.36)
  Study Visit 4* (only parental portion of ACT collected: Range 0-15) - Month 7: number analyzed (Participants) | 32 | 16 | 29
  Study Visit 4* (only parental portion of ACT collected: Range 0-15) - Month 7 | 2.29 (0.62) | 2.33 (0.86) | 2.36 (0.72)
  Study Visit 5* (only parental portion of ACT collected: Range 0-15) - Month 12: number analyzed (Participants) | 30 | 14 | 29
  Study Visit 5* (only parental portion of ACT collected: Range 0-15) - Month 12 | 1.75 (0.61) | 2.41 (0.71) | 1.74 (0.79)

4. Secondary Outcome: Number of Asthma-related Emergency Room Visits, Hospitalizations and Oral Steroid Courses
Description: Calculate and compare the number of asthma-related emergency room visits, hospitalizations and oral steroid courses between study arms.
Time Frame: 12 months
Population: The oral steroid course outcome was a secondary outcome added when we expanded inclusion criteria during the Coronavirus pandemic, so it is only reported for a proportion of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Incentives, Plus Reminders & Feedback (IRF) | Arm 2: Reminders & Feedback ONLY | Arm 3 (Control)
Number analyzed (Participants) | 38 | 21 | 40
Participants
  0 hospitalizations | 32 | 17 | 34
  1 hospitalization | 5 | 3 | 5
  2 hospitalizations | 1 | 1 | 0
  3 hospitalizations | 0 | 0 | 1
  0 emergency department visits | 31 | 14 | 27
  1 emergency department visit | 4 | 6 | 8
  2 emergency department visits | 3 | 0 | 2
  3 emergency department visits | 0 | 1 | 3
  0 oral steroid courses: number analyzed (Participants) | 30 | 13 | 25
  0 oral steroid courses | 21 | 4 | 13
  1 oral steroid course: number analyzed (Participants) | 30 | 13 | 25
  1 oral steroid course | 6 | 4 | 8
  2 oral steroid courses: number analyzed (Participants) | 30 | 13 | 25
  2 oral steroid courses | 1 | 3 | 1
  3 oral steroid courses: number analyzed (Participants) | 30 | 13 | 25
  3 oral steroid courses | 2 | 1 | 2
  4 oral steroid courses: number analyzed (Participants) | 30 | 13 | 25
  4 oral steroid courses | 0 | 0 | 1
  5 or more oral steroid courses: number analyzed (Participants) | 30 | 13 | 25
  5 or more oral steroid courses | 0 | 1 | 0

5. Secondary Outcome: Healthcare Costs of Utilization
Description: Calculate the costs associated with emergency room utilization, hospital utilization and oral steroid course prescriptions between study arms.
Time Frame: 12 months
Population: This secondary outcome will not be analyzed because this data was not collected for reasons related to the onset of the COVID-19 pandemic.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entirety of the participant's study period (12 months).
Description: Adverse events were only analyzed for the children involved in this study. The numbers differ with the number of individuals at risk for an adverse event due to participants that were lost to follow up, meaning that the participant had less than 14 days of electronic monitoring data following randomization, removing them from the study.
Arm/Group | Arm 1: Incentives, Plus Reminders & Feedback (IRF) | Arm 2: Reminders & Feedback ONLY | Arm 3 (Control)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/21 | 0/40
Serious Adverse Events (participants affected / at risk) | 6/38 | 4/21 | 6/40
Other Adverse Events (participants affected / at risk) | 17/38 | 13/21 | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Incentives, Plus Reminders & Feedback (IRF) (N=38) | Arm 2: Reminders & Feedback ONLY (N=21) | Arm 3 (Control) (N=40)
Asthma Exacerbation or Increased Asthma Symptoms (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Risk for Neurologic Deterioration (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Incentives, Plus Reminders & Feedback (IRF) (N=38) | Arm 2: Reminders & Feedback ONLY (N=21) | Arm 3 (Control) (N=40)
Asthma Exacerbation or Increased Asthma Symptoms (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 13
Joint/Extremity Pain or Fracture (Injury, poisoning and procedural complications) | 4 | 2 | 4
Hordeolum Externum (Infections and infestations) | 0 | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Otitis Externa (Infections and infestations) | 0 | 1 | 0
Seizures (Nervous system disorders) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 1
Concerns for glass ingestion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Flu (Infections and infestations) | 0 | 0 | 1
Balantitis Xerotica Obliterans (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tooth Pain/Dental Cavities (General disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
(1) The study included no "real world" control comparison group. Active control received electronic inhaler sensors with linked smartphone application which tracked medication usage and notified participants when usage changed. (2) The study had a relatively small sample size, though sufficiently powered to detect a difference between arm 1 (IRF) and arm 3 (active control). (3) The child portion of the Child Asthma Control Test (cACT, secondary outcome) was not completed at each study visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT03907410/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03907410/ICF_001.pdf